CLINICAL TRIAL: NCT05752760
Title: Impact of Lactobacillus Plantarum 299v Probiotic Supplementation on Vascular Function and Exercise Capacity in Chronic Heart Failure With Reduced and Preserved Ejection Fraction.
Brief Title: Pilot Study Lp299v Supplementation in Chronic Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Advancing a Healthier Wisconsin (Unknown)
Responsible Party: Principal Investigator, Michael E. Widlansky, MD, MPH, FACC, FAHA, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 45284
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure, Systolic; Heart Failure With Preserved Ejection Fraction; Heart Failure, Diastolic
Keywords: Endothelial Function; Microbiome; Heart Failure; Ejection Fraction
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lp299v (Experimental): Subjects will consume 20 billion colony forming units of Lp299v (2 capsules) once daily for 12 weeks.
  Interventions: Other: Lactobacillus Plantarum 299v Freeze Dried Capsule
- Placebo Control (Placebo Comparator): Subjects will consume potato starch (2 capsules) once daily for 12 weeks.
  Interventions: Other: Freeze Dried Potato Starch Capsule

INTERVENTIONS:
Other: Lactobacillus Plantarum 299v Freeze Dried Capsule — The intervention is a probiotic lactobacillus that is contained in food products in the US
  Arms: Lp299v
Other: Freeze Dried Potato Starch Capsule — The intervention is potato starch that is freeze dried designed to mimic the lp299v capsule.
  Arms: Placebo Control

SUMMARY:
The goal of this study is to determine the impact of 12 weeks of Lp299v supplementation (20 million cfu/day vs. placebo) on exercise capacity, circulating biomarkers of cardiac remodeling, quality of life, and vascular endothelial function in humans with heart failure and reduced ejection fraction (HFrEF) and heart failure with preserved ejection fraction (HFpEF) who have evidence of residual inflammation based on an elevated C-reactive protein level. This will be done in the setting of a randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Heart failure (HF) has significant morbidity and mortality and is one of the leading causes of hospital admissions in the United States. In 2017, almost 1 million people were affected and responsible for 1.2 million hospitalizations in the United States alone. Prognosis is poor for patients with HF despite significant medical therapy regimens and device therapy. Worldwide, mortality is as high as 17% during initial hospitalization, as high as 45% within one year of admission, and greater than 50% within five years. According to the Wisconsin Department of Health Services, mortality rates for HF have been increasing in the state since 1980. Wisconsin also consistently had higher rates of HF compared to the remaining states.

Emerging data suggest targeting the gut microbiota in HF could be a safe and effective alternative for mitigating inflammation. HF patients have increased systemic circulating endotoxins and lipopolysaccharides due to impaired gut-barrier function, secondary to gut congestion and reduced cardiac output, which drives systemic inflammation. The gut flora of patients with HF also includes more pathogenic bacteria species (candida, campylobacter, shigella, and yersinia) compared to patients with normal heart function.

Previous studies by the lab showed that supplementation of 20 billion cfu/day of Lactobacillus plantarum 299v (Lp299v) probiotic decreases systemic inflammation in men with stable coronary artery disease (CAD), and also improves vascular endothelial function (measured by endothelium-dependent vasodilation in the brachial artery and by nitric-oxide dependent vasodilation of resistance arterioles from CAD patients). The investigators have shown that there are significantly decreased levels of IL-8, IL-12 and Leptin in Lp299v-supplemented patients with CAD. Leptin is known to increase IL-6 (which drives increased C-reactive protein expression), IL-8, IL-12 and TNF-α levels, all which activate pro-inflammatory immune responses leading to vasoconstriction and vascular stiffness. Further, our data suggests Lp299v has a significant, favorable anti-inflammatory effect on signaling pathways (NLRP3, IL-6, IL-1β) shown to be important to chronic inflammation in heart failure.

Therefore, the investigators plan to perform a pilot study targeting the gut microbiota of patients with HF with oral supplementation with 20 billion cfu/day of Lp299 and determine if Lp299v improves peak oxygen consumption (measured by VO2 max testing), endothelial function (measured by brachial artery flow-mediated dilation), and vascular stiffness (measured by peak wave velocity). We plan to test the hypothesis that Lp299v will improve these measures in the setting of a randomized, double-blind, placebo-controlled clinical trial of 20 subjects. The investigators will additionally test if Lp299v supplementation improves circulating biomarkers of inflammation and cardiac remodeling in chronic heart failure, as well as if it improves the quality of life in patients using the Minnesota Living with Heart Failure Questionnaire and the Kansas City Cardiomyopathy Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-89 years old
* Clinical diagnosis of Congestive Heart Failure (CHF) in the six months prior to enrollment along with an echocardiogram documenting systolic dysfunction with ejection fraction ≤40%
* Clinical diagnosis of CHF in the six months prior to enrollment along with an echocardiogram documenting diastolic dysfunction with an ejection fraction ≥50%, and a H2FpEFF score of ≥6
* New York Heart Association (NYHA) Class II-IIID heart failure symptoms with either ischemic or non-ischemic etiology OR similar diagnosis with congestive heart failure (CHF) along with an echocardiogram documenting an LV ejection fraction of 50% or more with similar NYHA classification as those with LVEF of 40% or less
* Evidence of systemic inflammation at baseline (C-reactive protein ≥ 2 mg/L at the time of screening)

Exclusion Criteria:

* Heart failure due to severe valve disease such as Aortic Stenosis, Mitral Regurgitation, or Mitral Stenosis
* Cancer besides non-melanoma skin carcinomas or localized prostate and breast cancer at the time of enrollment with life expectancy <1 year
* Lung disease such as Chronic Obstructive Pulmonary Disease (COPD), emphysema, or Pulmonary fibrosis
* Active inflammatory disease or infectious disease at the time of enrollment
* Current treatment (or use within the past 14 days) of steroids or anti-inflammatory treatments (excluding non-steroidal anti-inflammatory medications or steroids used solely for IV contrast dye allergy)
* Chronic Kidney Disease with eGFR ≤ 30 mL/min
* Hepatic Failure (Child's Class B or C)
* Patients with Gastrointestinal (GI) tract illness such as short gut syndrome, inflammatory bowel disease, or an ileostomy, such that probiotic absorption would be altered
* Anticipated need for cardiac surgery during the projected study period for the subject
* Pregnancy
* Patients who are receiving Vitamin K antagonists such as Coumadin or Warfarin
* Neutropenia (Absolute Neutrophil Count (ANC) < 1800/mm3)
* Inability to give informed consent or follow the study protocol
* On antibiotics at the time of enrollment or within one month of enrollment
* Currently taking a Lactobacillus based probiotic as an outpatient at the time of enrollment
* Patients who are unable to walk on treadmill or use a bicycle to participate in exercise testing
* Allergy to Lp299v probiotic supplement

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Oxygen Consumption (VO2Max) | 12 weeks
  This is a measurement of exercise capacity
Brachial Artery Flow Mediated Dilation (FMD%) | 12 weeks
  This is a measurement of endothelial function in the brachial artery
Carotid-Femoral Pulse Wave Velocity (cfPWV) | 12 weeks
  Measurement of vascular stiffness

SECONDARY OUTCOMES:
Brachial Artery Absolute Flow Mediated Dilation (FMDmm) | 12 weeks
  This is a measurement of endothelial function in the brachial artery
Resting shear stress of brachial artery | 12 weeks
  This is a measurement of vascular stiffness
Resting velocity | 12 weeks
  This is a measurement of vascular stiffness
Change in serum Soluble Suppression Tumorigenesis (SST2) | 12 weeks
  This measures cardiac fibrosis
Peak flow velocity | 12 weeks
  This is a measurement of vascular stiffness
Peak Hyperemic Shear Stress of Brachial Artery | 12 weeks
  This is a measurement of vascular stiffness
Change in Galectin-3 | 12 weeks
  This measures cardiac fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Widlansky, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Within 1 year of completion of all studies procedures

REFERENCES:
- [Background] Agarwal MA, Fonarow GC, Ziaeian B. National Trends in Heart Failure Hospitalizations and Readmissions From 2010 to 2017. JAMA Cardiol. 2021 Aug 1;6(8):952-956. doi: 10.1001/jamacardio.2020.7472. PMID 33566058
- [Background] Dick SA, Epelman S. Chronic Heart Failure and Inflammation: What Do We Really Know? Circ Res. 2016 Jun 24;119(1):159-76. doi: 10.1161/CIRCRESAHA.116.308030. PMID 27340274
- [Background] Wisconsin Heart Disease and Stroke Prevention Program, February 2010. www.dhs.wisconsin.gov/publications/p0/p00146.pdf
- [Background] Pasini E, Aquilani R, Testa C, Baiardi P, Angioletti S, Boschi F, Verri M, Dioguardi F. Pathogenic Gut Flora in Patients With Chronic Heart Failure. JACC Heart Fail. 2016 Mar;4(3):220-7. doi: 10.1016/j.jchf.2015.10.009. Epub 2015 Dec 9. PMID 26682791
- [Background] Hofeld BC, Puppala VK, Tyagi S, Ahn KW, Anger A, Jia S, Salzman NH, Hessner MJ, Widlansky ME. Lactobacillus plantarum 299v probiotic supplementation in men with stable coronary artery disease suppresses systemic inflammation. Sci Rep. 2021 Feb 17;11(1):3972. doi: 10.1038/s41598-021-83252-7. PMID 33597583
- [Background] Iikuni N, Lam QL, Lu L, Matarese G, La Cava A. Leptin and Inflammation. Curr Immunol Rev. 2008 May 1;4(2):70-79. doi: 10.2174/157339508784325046. PMID 20198122
- [Background] Santos-Alvarez J, Goberna R, Sanchez-Margalet V. Human leptin stimulates proliferation and activation of human circulating monocytes. Cell Immunol. 1999 May 25;194(1):6-11. doi: 10.1006/cimm.1999.1490. PMID 10357875
- [Background] Spertus, J., Kansas City Cardiomyopathy Questionnaire MDDT decision summary. <fda.gov>
- [Background] Thomas, R, Cohn, J., Minnesota Living with Heart Failure Questionnaire <license.umn.edu/product/minnesota-living-with-heart-fialure-questionnaire-mlhfq>